CLINICAL TRIAL: NCT03574051
Title: Distinct Shifts in the Microbiota Are Associated With Iodine-131 Therapy and Hypothyroidism
Brief Title: the Microbiota Are Associated With Iodine-131 Therapy and Hypothyroidism
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yunwei Wei 2018 -05-21
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-05

CONDITIONS: Microbiota
Keywords: oral microbiota; 16S rRNA gene; thyroid cancer; iodine 131 treatment; fecal microbiota; radiotherapy
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Probiotic (Experimental): Taking probiotics containing Bifidobacterium infantis, Lactobacillus acidophilus and Enterococcus faecalis for 30 days
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — Evaluate probiotics for preventing adverse effects of hypothyroidism and improvement of side effects caused by 131I treatment
  Other Names: Complex-probiotic-preparation

SUMMARY:
Thyroid cancer is a common neck malignancy. Currently, total thyroidectomy or subtotal thyroidectomy is the main method for the treatment of thyroid cancer patients. However, some thyroid cancer may still have residual thyroid tissue after operation. Therefore, in the differentiated thyroid In the treatment of cancer, iodine 131 treatment is mainly used because iodine 131 can emit high-energy beta rays, destroying the residual tissue of thyroid cancer and achieving good therapeutic goals. However, in the treatment of iodine-131, certain salivary glands are inevitably damaged, and the patient will have dry mouth symptoms. After the same treatment with iodine-131, some patients will experience gastrointestinal reactions such as nausea and vomiting. The therapeutic efficacy of iodine-131 depends on the lesion's uptake of iodine-131, which requires an increase in serum TSH levels. All patients in this study had stopped taking thyroid hormone for 3-4 weeks before iodine 131 treatment, making serum The TSH level is greater than 30 mU/L. At this time, the patient is in hypothyroidism. People with hypothyroidism experience dry mouth, dry skin, constipation, pain, cold, poor memory, depression, and weight gain. Many studies have pointed out that some cancer treatments, such as chemotherapy and radiotherapy, also have an impact on the microbial flora. However, studies on the relationship between microecology, hypothyroidism and iodine-131 treatment, probiotics in the prevention of hypothyroidism and iodine-131 treatment The link between the effects of side effects remains unclear. Therefore, the team will conduct a correlation study between microbes and hypothyroidism, iodine-131 treatment.

DETAILED DESCRIPTION:
Thyroid cancer is a common neck malignancy and it mainly affects thyroid follicular cells or parafollicular cells. Thyroid cancer in various tumors in the body, the ratio can reach 1.2% to 2.3%. Thyroid cancer can be divided into differentiated thyroid cancer, squamous cell carcinoma, undifferentiated carcinoma, and medullary carcinoma, among which the incidence of differentiated thyroid carcinoma is more than 90%. At present, total thyroidectomy or subtotal thyroidectomy is the main method for the treatment of thyroid cancer patients, but some thyroid cancer may still have residual thyroid tissue after operation. Therefore, in the treatment of differentiated thyroid cancer, iodine 131 is mainly used. Treatment, because iodine 131 can emit high-energy beta rays, destroying the residual tissue of thyroid cancer, to achieve good therapeutic purposes. However, due to the presence of sodium iodine symporter in salivary glands and thyroid, it is inevitable that certain salivary glands will be damaged in the treatment of iodine 131, and patients will have dry mouth symptoms. Some patients with nausea 131 will also experience nausea and vomiting. Gastrointestinal reaction. Iodine 131 treatment is divided into two steps: 1 removal of residual thyroid tissue; 2 removal of cancer lesions and metastases. The curative effect of 131I depends on the lesion's uptake of iodine-131, which requires an increase in serum TSH levels. All patients in this study had stopped taking thyroid hormone for 3 to 4 weeks before iodine-131 treatment. The TSH level is greater than 30 mU/L. At this time, the patient is in hypothyroidism. People with hypothyroidism experience dry mouth, dry skin, constipation, pain, cold, poor memory, depression, and weight gain. Many studies have pointed out that some cancer treatments, such as chemotherapy and radiotherapy, also have an impact on the microbial flora. However, studies on the relationship between microecology, hypothyroidism and iodine-131 treatment, probiotics in the prevention of hypothyroidism and iodine-131 treatment The link between the effects of side effects remains unclear. Therefore, the team will conduct a correlation study between microbes and hypothyroidism, iodine-131 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old, 65 years old, male and female;
* Histologically confirmed differentiated thyroid cancer;
* After total thyroidectomy, patients who have undergone 131I therapy for the second time or more after recurrence or regional lymph node metastasis after 131I treatment for the first time are required. Or after the first 131I treatment, patients with differentiated thyroid who were treated with 131I for more than 3 months.

Exclusion Criteria:

* Use of various antibiotics within three months;
* Having a history of alcoholism for more than 2 years and a history of smoking throughout the year;
* pregnancy or lactation;
* having oral, respiratory and gastrointestinal diseases;
* has a variety of metabolic diseases, such as obesity, hypertension, diabetes, stones, various liver diseases, etc.;
* having other autoimmune diseases such as rheumatoid arthritis, ankylosing spondylitis, inflammatory bowel disease, etc.;
* History of gastrointestinal surgery or other recent surgical history;
* Has a family history of genetic disease, mental illness, etc.;
* Research subjects are participating in other research topics;
* The researchers believe that other reasons are not suitable for continuing clinical trials;
* Undifferentiated thyroid cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients with improved side effects | 4 weeks
  Improved side-effects in patients, such as reduced diarrhea and improved dry mouth symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yunwei Wei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verburg FA, Hanscheid H, Luster M. Radioactive iodine (RAI) therapy for metastatic differentiated thyroid cancer. Best Pract Res Clin Endocrinol Metab. 2017 Jun;31(3):279-290. doi: 10.1016/j.beem.2017.04.010. Epub 2017 May 9. PMID 28911724
- [Background] Ciorba MA, Riehl TE, Rao MS, Moon C, Ee X, Nava GM, Walker MR, Marinshaw JM, Stappenbeck TS, Stenson WF. Lactobacillus probiotic protects intestinal epithelium from radiation injury in a TLR-2/cyclo-oxygenase-2-dependent manner. Gut. 2012 Jun;61(6):829-38. doi: 10.1136/gutjnl-2011-300367. Epub 2011 Oct 24. PMID 22027478
- [Background] Linn YH, Thu KK, Win NHH. Effect of Probiotics for the Prevention of Acute Radiation-Induced Diarrhoea Among Cervical Cancer Patients: a Randomized Double-Blind Placebo-Controlled Study. Probiotics Antimicrob Proteins. 2019 Jun;11(2):638-647. doi: 10.1007/s12602-018-9408-9. PMID 29550911
- [Derived] Lin B, Zhao F, Liu Y, Wu X, Feng J, Jin X, Yan W, Guo X, Shi S, Li Z, Liu L, Chen H, Wang H, Wang S, Lu Y, Wei Y. Randomized Clinical Trial: Probiotics Alleviated Oral-Gut Microbiota Dysbiosis and Thyroid Hormone Withdrawal-Related Complications in Thyroid Cancer Patients Before Radioiodine Therapy Following Thyroidectomy. Front Endocrinol (Lausanne). 2022 Mar 8;13:834674. doi: 10.3389/fendo.2022.834674. eCollection 2022. PMID 35350100